CLINICAL TRIAL: NCT05087329
Title: Mindfulness Practice in Pregnancy As an Intervention to Decrease Prenatal Stress During the COVID-19 Pandemic
Acronym: CALMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: additional studies in this specific population made continuing with RCT unnecessary so became a part of clinical care
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kirstin Leitner, Assitant Professor of Obstetrics and Gynecology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 843962
Record Dates: First submitted 2021-10-19; First posted 2021-10-21 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-02

CONDITIONS: Prenatal Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Mindfulness intervention (Experimental): Four weekly group Zoom webinars with a 15-20 minute pre-recorded meditation
  Interventions: Behavioral: Virtual Mindfulness Meditation
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Virtual Mindfulness Meditation — Four week virtual mindfulness meditation course composed of four weekly group Zoom webinars during which participants will listen to a 15-20 minute pre-recorded meditation, facilitated by a study provider
  Arms: Virtual Mindfulness intervention

SUMMARY:
The purpose of the study is to examine whether a simple mindfulness intervention conducted via a virtual platform can reduce stress among pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 16w0d-26w6d gestation with a single gestation who have had a confirmed dating ultrasound

   a. Only women with singleton gestations will be included because multiple gestation pregnancies introduce additional levels of stress and introduce confounding variables for the adverse composite pregnancy outcome that will be measured. As this is a study of pregnant patients, only women are included.
2. English speaking

   a. The mindfulness meditation trainings have been scripted and recorded in English. Thus, to understand the recordings and participate in the courses it is necessary for all participants to speak English.
3. Regular internet access through either phone, tablet or computer. a. Mindfulness meditations are administered via Zoom webinars so internet access is required. A proxy for internet access during recruitment will be confirmed by the inclusion of an email address in the electronic medical record (EMR).

Exclusion Criteria:

1. Multiple gestations. This has been chosen as an exclusion criteria to limit confounding variables for the secondary outcome of composite adverse pregnancy events.
2. Age < 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Decrease in Maternal Stress | 6 to 8 weeks
  Change in score on Perceived Stress Scale (PSS)

SECONDARY OUTCOMES:
Composite score of maternal morbidity/pregnancy outcomes | 6 to 8 weeks post-delivery
Change in score on Edinburgh Postnatal Depression Scale | change between score at time of delivery and 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadephia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No